CLINICAL TRIAL: NCT00600197
Title: The Effectiveness of Biopsychosocial Education on Quality of Life and Disability of Individuals Suffering From Chronic Low Back Pain
Brief Title: Biopsychosocial Education and Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sedigheh Sadat Tavafian, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 86-03-41-5465
Record Dates: First submitted 2008-01-13; First posted 2008-01-24 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Back school (Experimental): a kind of educational program for low back pain
  Interventions: Behavioral: back school
- back school (Experimental)
  Interventions: Behavioral: back school

INTERVENTIONS:
Behavioral: back school — A kind of educational program for low back pain

SUMMARY:
The purpose of this study is to examine whether the biopsychosocial educational program could improve patients' health-related quality of life at 3-6-12-18-24-30 and 36 - month follow up.

DETAILED DESCRIPTION:
Little information exists on biopsychosocial educational program as a multidimensional and interdisciplinary program in which Quality Of Life is as an outcome measure. Thus this educational Program designed in this study is a an outpatient program that used a health education approach to empower participants through a process of assessment, education and skill building in three dimensions of physical,mental and social that leading to improved quality of life. The purpose of this study was to examine to what extent this educational Program could improve low back pain patients' HRQOL.

ELIGIBILITY:
Inclusion Criteria:

* Low Back Pain lasting more than 12 weeks with or without pain radiating to the legs.
* age 18-70 years.

Exclusion Criteria:

* Osteoporosis
* Newly operation on the back up to 2 years before the beginning of the study
* Fresh vertebral fracture
* Malignancy
* Infection in the back
* spondylolisthesis
* Problem in understanding Farsi Language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-04 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
SF-36, Roland Morris Disability Questionnaire, Quebec back pain disability | before intervention

SECONDARY OUTCOMES:
SF-36,Roland Morris Disability Questionnaire, Quebec back pain disability | 3-6-12-18-24-30-36 month after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Re Jamshidi, MD, Study Chair — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Tavafian SS, Jamshidi AR, Mohammad K. Treatment of low back pain: randomized clinical trial comparing a multidisciplinary group-based rehabilitation program with oral drug treatment up to 12 months. Int J Rheum Dis. 2014 Feb;17(2):159-64. doi: 10.1111/1756-185X.12116. Epub 2013 Jun 21. PMID 24576271